CLINICAL TRIAL: NCT01271400
Title: Use of the LANDA Embryo Freezing Technique to Validate Frozen Embryo Transfer Success Rates
Brief Title: LANDA Embryo Freezing Technique.
Acronym: Freezing
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West Coast Fertility Centers (Other)
Responsible Party: Principal Investigator, David G. Diaz, MD, Medical Director, West Coast Fertility Centers
Other Study IDs: 2010-1
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Primary Infertility; Secondary Infertility; Genital Diseases, Male; Genital Diseases, Female
Keywords: Infertility treatments; Frozen embryo transfers (FET).; IVF.; ART.; Cryopreservation; Slow-Freeze; Freeze / thaw survival rates; Blastocyst formation; Pregnancy
MeSH Terms: conditions — Genital Diseases, Male; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to track the outcome from the patients who had embryo cryopreservation as part of their Advanced Reproductive Technology (ART) treatment at West Coast Fertility Centers.

DETAILED DESCRIPTION:
Over the past several decades, considerable effort has been expended toward the successful cryopreservation of various human cells. While attempts at cryopreservation have been directed at different tissue types, one of the most vigorously pursued targets has been reproductive tissue. Historically, cryopreservation of human sperm has existed for several decades. The earliest reports of pregnancies (Trounson et al., 1983) and births (Zeilmaker et al., 1984) from the cryopreservation of human embryos occurred in the early 1980s. Presently, the freezing and storage of human embryos following in vitro fertilization (IVF) is standard practice at most fertility clinics. In 2003, the CDC Assisted Reproductive Technology success rates report stated that 4,246 live births occurred out of 17,517 non-donor frozen embryo cycles.

Embryo cryopreservation has been a routine component of clinical IVF programs for more than 2 decades but has a relatively poor outcome in terms of post-thaw survival and pregnancy rates in a majority of IVF programs. Efficient embryo cryopreservation has several advantages. It helps to reduce costs and increases cumulative pregnancy rates. It can also help in cases of IVF cycles where embryos are not transferred due to ovarian hyper stimulation syndrome. It is also useful when technical difficulties are encountered at the time of an embryo transfer procedure.

One of the major concerns in IVF is high-order multiple pregnancies, which result from the transfer of multiple embryos in a given cycle. In the last 5 years, improved stimulation protocols, advances in culture and laboratory systems, and better identification of viable embryos have enhanced the success rates of IVF. During the same period, some clinics have started the practice of transferring two embryos to reduce multiple pregnancy rates without compromising overall pregnancy rates.

Furthermore, in recent years some European countries, particularly the Scandinavian countries, have taken a lead in performing elective single-embryo transfers and have achieved acceptable pregnancy rates. This trend is spreading to other countries. This can result in surplus embryos being available for freezing. With the application of ICSI, even patients aged 40 years or older may have embryos to freeze.

Review of the current literature reveals modest post-thaw embryo survival, implantation, and pregnancy rates. Post-thaw survival rates vary from 50% to 80% for different embryo stages. Implantation and pregnancy rates have varied from 3% to 15% and 15% to 25% respectively, which is approximately half of the rates achieved for fresh embryo transfers.

To improve the outcome of frozen ET cycles, we modified various steps of our standard cryopreservation protocol. In a pilot study on arrested and fragmented embryos (grades 3 and 4), we achieved post-thaw survival rates of 92%, having all blastomeres intact. Encouraged by the post-thaw survival of these embryos; we propose using this modified protocol in our frozen embryo transfer program.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion into this study, each subject must satisfy the following criteria:

  1. Infertile women whose physician has recommended IVF and who agree to cryopreserve surplus embryos.
  2. Cancer patients who wish to preserve their fertility prior to cancer treatments.
  3. Recipients who wish to use frozen donor embryos.
  4. A male partner whose semen analysis meets the clinic criteria for ICSI. Use of donor sperm is also acceptable.
  5. Be willing and able to comply with the protocol for the duration of the study.
  6. Have voluntarily provided written informed consent under WIRB.

Exclusion Criteria:

* A patient may NOT be entered into the study if she presents with ANY of the following criteria:

  1. Clinically significant systemic disease.
  2. Known endometriosis Grade III - IV (ASRM classification).
  3. Any previous cycle indicating a low response to gonadotropin stimulation (defined as retrieval of < 10 eggs at retrieval)
  4. Three or more previous ART cycles without a clinical pregnancy
  5. Abnormal, undiagnosed, gynecological bleeding.
  6. Previous ovarian surgery
  7. Known allergy or hypersensitivity to recombinant gonadotropin preparations or any other study-related medications.
  8. Verifiable substance abuse.
  9. Simultaneous participation in another study protocol.
  10. Current smoker.
  11. An extrauterine pregnancy within the last 3 months before OCP treatment commences.

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertility patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Freeze/Thawed survival rates | When embryos thawed initiate
  * Freeze / thaw survival rates
  * Blastocyst formation rates
  * Pregnancy rate.

CONTACTS AND LOCATIONS:
Overall Officials: David G. Diaz, M.D., Principal Investigator — West Coast Fertility Centers
Locations (1):
- West Coast Fertility Centers, Fountain Valley, California, United States